CLINICAL TRIAL: NCT01482767
Title: A Prospective, Phase III, Open-Label Study of Boceprevir, Pegylated-Interferon Alfa 2b and Ribavirin in HCV/HIV Coinfected Subjects
Brief Title: Evaluating the Effectiveness of Boceprevir, Pegylated-Interferon Alfa 2b and Ribavirin in Treating Hepatitis C Virus (HCV) Infection in Adults With HIV and HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5294 (BIRTH); 11774 (Registry Identifier: DAIDS ES); ACTG 5294; BIRTH
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Results first posted 2016-05-10 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2016-06

CONDITIONS: HIV Infections; Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HCV Treatment-Naive (Group A) (Experimental): Participants were prescribed a lead-in with PEG-IFN and RBV for 4 weeks. After the lead-in, BOC was added. Cirrhotic participants received 44 weeks of triple therapy (BOC+PEG-IFN+RBV). Among non-cirrhotics, the Week 8 HCV RNA was used to determine total duration of therapy. Those who had undetectable HCV RNA at Week 8 completed therapy at Week 28. Those with detectable HCV RNA at Week 8 received 32 weeks of triple therapy followed by 12 additional weeks of PEG-IFN+RBV.
  Interventions: Drug: Pegylated-Interferon Alfa 2b (PEG-IFN); Drug: Ribavirin (RBV); Drug: Boceprevir (BOC)
- HCV Treatment-Experienced (Group B) (Experimental): Participants were prescribed a lead-in with PEG-IFN and RBV for 4 weeks. After the lead-in, BOC was added. Cirrhotic participants received 44 weeks of triple therapy (BOC+PEG-IFN+RBV), and non-cirrhotics received 32 weeks of triple therapy followed by 12 additional weeks of PEG-IFN+RBV.
  Interventions: Drug: Pegylated-Interferon Alfa 2b (PEG-IFN); Drug: Ribavirin (RBV); Drug: Boceprevir (BOC)

INTERVENTIONS:
Drug: Pegylated-Interferon Alfa 2b (PEG-IFN) — 1.5 mcg/kg subcutaneously (SC) once a week (based on participant's weight at entry) for up to 48 weeks depending on cirrhosis status and, in Group A, Week 8 HCV viral response.
Drug: Ribavirin (RBV) — 800-1400 mg orally per day with food (based on participant's weight at entry) for up to 48 weeks depending on cirrhosis status and, in Group A, Week 8 HCV viral response.
Drug: Boceprevir (BOC) — 800 mg orally every 8 hours with food from Week 5 to up to Week 48 depending on cirrhosis status and, in Group A, Week 8 HCV viral response

SUMMARY:
Hepatitis C virus (HCV) infection is a leading cause of death and illness in people with HIV-1. At the time the study was designed, the standard treatment for people with HIV-1 and HCV coinfection included two drugs: pegylated-interferon alfa 2b (PEG-IFN) and ribavirin (RBV). The purpose of this study was to evaluate the effectiveness of giving boceprevir (BOC) together with standard treatment in treating HCV infection in people with HIV-1 and HCV coinfection.

DETAILED DESCRIPTION:
For HIV-1-infected individuals, HCV infection is a leading cause of morbidity and mortality, and the prevalence of HCV infection is higher among those infected with HIV-1. At the time the study was designed, the standard-of-care (SOC) therapy for HCV infection was treatment with both PEG-IFN and RBV. This therapy is 40%-45% effective in patients with HCV infection but is significantly less effective in patients with both HCV and HIV-1 (Shire et al. J Viral Hepat., 2007). The purpose of this study was to evaluate the effectiveness of adding BOC (Kwo et al. Lancet, 2010), an HCV protease inhibitor, to SOC therapy in treating HCV infection (genotype 1) in HCV/HIV-1-coinfected adults.

Participants were enrolled into one of two groups based on previous HCV treatment experience.

1. Group A: HCV treatment-naive participants who had never received treatment with PEG-IFN or experimental agents used to treat HCV, with or without RBV (N=170, refer to the note below).
2. Group B: HCV treatment-experienced participants who had received any treatment with standard interferon or with PEG-IFN with or without RBV, provided the last dose of treatment was 90 days or more before study entry (N=140, refer to the note below).

Note: The team correspondence with the FDA led to an amendment to close enrollment in December 2013, prior to the target sample sizes of 170 in Group A and 140 in Group B, as the study power could be lowered while still meeting the key study objectives.

All participants had to be on stable antiretroviral therapy (ART) for at least 8 weeks prior to study entry using a dual nucleos(t)ide reverse transcriptase inhibitor (NRTI) backbone plus one of the following: efavirenz (EFV), raltegravir (RAL), lopinavir (LPV)/ritonavir (RTV) 400/100 mg twice daily, atazanavir (ATV)/RTV, darunavir (DRV)/RTV 600/100 mg twice daily OR must not have received any ART for at least 4 weeks immediately prior to entry. Participation in this study lasted approximately 72 weeks.

HCV treatment-naive participants (Group A) were treated with PEG-IFN and RBV for 4 weeks (lead-in). Then BOC was added to the treatment regimen (triple therapy). Cirrhotic participants received 44 weeks of triple therapy. Among non-cirrhotics, the Week 8 HCV RNA was used to determine total duration of therapy. Those who had undetectable HCV RNA at Week 8 completed therapy at Week 28. Those with detectable HCV RNA at Week 8 received 32 weeks of triple therapy followed by 12 additional weeks of double-drug therapy with PEG-IFN/RBV. HCV treatment-experienced participants (Group B) also had a lead-in followed by 32 weeks of triple therapy and 12 weeks of PEG-IFN/RBV double therapy if non-cirrhotic, or by 44 weeks of triple therapy if cirrhotic.

Treatment was to be discontinued due to HCV virologic failure if:

1. HCV RNA ≥100 IU/mL at Week 12,
2. detectable HCV RNA at Week 24, or
3. confirmed HCV RNA >1000 IU/mL any time after Week 12.

Undetectable HCV RNA was defined as below the lower limit of quantification (LLOQ) and target not detected (TND) by Roche COBAS® TaqMan® HCV Test v2.0.

Study visits were scheduled at screening and at Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24 and 28 for both study groups. Group A participants who completed treatment at Week 28 had further study visits at Weeks 40, 52, 60, and 72. Participants who were prescribed 48-weeks of therapy (Group A and Group B) had further study visits at Weeks 32, 36, 40, 44, 48, 60, and 72. At each visit, a physical examination and blood collection were conducted. Participants also completed an HCV treatment adherence questionnaire. Select visits included urine collection and pregnancy testing (for women of reproductive potential). Plasma, serum, and peripheral blood mononuclear cells (PBMCs) were be stored for use in future studies. After experiencing HCV virologic failure as defined above or premature treatment discontinuation due to safety or other reasons, participants were followed on a separate schedule of events with visits every 12 weeks from Week 24 to 72. The evaluations at these follow-up visits were limited to safety evaluations and stored plasma/serum sample collection.

The A5294 study consisted of single-arm evaluations to assess the efficacy of BOC added to PEG-IFN/RBV in the two study populations:

1. HCV treatment-naive participants (Group A)
2. HCV treatment-experienced participants (Group B).

The two study populations were addressed together in this single trial - rather than in two separate trials - mainly for administrative efficiency. The analyses were conducted separately for each Study Group. The study was not designed for comparison. The pooled summaries for Baseline Characteristics provided in the Results Section in this record were prepared solely for the ClinicalTrials.gov results submission.

ELIGIBILITY:
Inclusion Criteria (Groups A and B):

* Men and women 18 years of age or older
* Presence of chronic HCV infection, defined by presence of plasma or serum HCV RNA in a participant with HCV antibody for at least 180 days, two documented HCV RNA positive results greater than 180 days apart, or positive HCV RNA with biopsy demonstrating chronic hepatitis. More information on this criterion can be found in the protocol.
* Serum or plasma HCV RNA level 10,000 IU/mL or greater obtained within 42 days prior to study entry.
* Screening HCV genotype 1 performed within 6 months prior to study entry.
* Liver biopsy or HCV FibroSURE™ test within 104 weeks prior to study entry with interpretation consistent with chronic HCV infection. If a liver biopsy HCV FibroSURE™ test had not been performed within 104 weeks prior to study entry, then either a biopsy or HCV FibroSURE™ test must have been obtained prior to enrollment. The cut-off value for the FibroSURE™ test was 0.74, where greater than 0.74 was interpreted as cirrhosis. More information on this criterion can be found in the protocol.
* Alpha feto protein (AFP) levels less than 50. If 50 or greater, they must have had a liver imaging study (e.g., ultrasound, computed tomography [CT] scan, magnetic resonance imaging [MRI] showing no evidence of hepatocellular carcinoma.
* HIV-1 infection. More information on this criterion can be found in the protocol.
* Currently not on any antiretroviral therapy (ART) for at least 4 weeks immediately prior to entry or on stable ART for at least 8 weeks prior to study entry using a dual NRTI backbone PLUS one of the following: EFV, RAL, LPV/RTV 400/100 mg twice daily, ATV/RTV, DRV/RTV 600/100 mg twice daily. Breaks in therapy for a maximum of 14 days were allowed. Dose modifications or changes in drugs during the 8 weeks prior to study entry were permitted unless the change in drug was due to treatment failure. More information on this criterion can be found in the protocol.
* CD4+ T-cell count greater than 200 cells/mm^3 obtained within 42 days prior to study entry.
* For participants on ART, screening plasma HIV-1 RNA less than 50 copies/mL obtained within 42 days prior to study entry. For participants not on ART, plasma HIV-1 RNA less than 50,000 copies/mL obtained within 42 days prior to study entry.
* The following laboratory values within 42 days prior to entry:

  * Absolute neutrophil count (ANC) 1000/mm^3 or greater,
  * Hemoglobin greater than 12 g/dL for men and greater than 11 g/dL for women,
  * Platelet count greater than 80,000 per mm^3,
  * Creatinine less than 1.5 mg/dL,
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT), alkaline phosphatase (ALT)/serum glutamic pyruvic transaminaseless (SGPT) less than or equal to 10 x the upper limit of normal (ULN),
  * Direct bilirubin less than 1.5 mg/dL,
  * International normalized ratio (INR) less than 1.5,
  * Serum lipase less than or equal to 1.5 x ULN,
  * Thyroid stimulating hormone (TSH) within normal range, unless accompanied by thyroid profile consistent with normal thyroid function.
* For female participants of reproductive potential, a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL performed within 42 days prior to study entry. More information on this criterion can be found in the protocol.
* All participants must have agreed not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization).
* When participating in sexual activity that could lead to pregnancy, participants must have agreed to use at least two reliable methods of contraception simultaneously while receiving protocol-specified medications, and for 6 months after stopping the medications. Such methods include:

  * Condoms (male or female) with a spermicidal agent,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Tubal ligation.

More information on this criterion can be found in the protocol.

* Participants not of reproductive potential were eligible without requiring the use of contraceptives. More information on this criterion can be found in the protocol.
* Ability and willingness of participant to provide written informed consent.

Exclusion Criteria (Groups A and B):

* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
* Evidence of decompensated liver disease manifested by the presence of or history of ascites, variceal bleeding, or hepatic encephalopathy. If hepatic cirrhosis was determined by liver biopsy (Stage 4 Metavir or Stage 5, 6 Ishak) or by imaging, then participants had to be no more than Child-Pugh Class A and have a Child-Pugh-Turcotte (CPT) score of 6 or less. More information on this criterion can be found in the protocol.
* Other known causes of significant liver disease including chronic or acute hepatitis B, acute hepatitis A, hemochromatosis, or homozygote alpha-1 antitrypsin deficiency.
* Infection with any HCV genotype other than genotype 1, or mixed genotype infection.
* Uncontrolled or active depression or other psychiatric disorder such as untreated. Grade 3 psychiatric disorder or Grade 3 disorder not amenable to medical intervention that in the opinion of the site investigator might have precluded tolerability or safety of study requirements. Individuals with suicidal ideation or history of a suicidal attempt in the last 5 years prior to enrollment were excluded.
* History of uncontrolled seizure disorders.
* Serious illness including malignancy, active coronary artery disease within 24 weeks prior to study entry, or other chronic medical conditions that in the opinion of the site investigator may have precluded completion of the protocol.
* Presence of active or acute AIDS-defining opportunistic infections within 12 weeks prior to study entry. More information on this criterion can be found in the protocol.
* History of hemoglobinopathy (e.g., thalassemia) or any other cause of or tendency to hemolysis.
* History of major organ transplantation with an existing functional graft.
* History of autoimmune processes including Crohn's disease, ulcerative colitis, severe psoriasis, or rheumatoid arthritis that may be exacerbated by IFN use.
* Breastfeeding.
* Male participants with pregnant sexual partner.
* Use of granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 14 days prior to study entry.
* Use of systemic corticosteroids, lovastatin, simvastatin, interferon gamma, tumor necrosis factor(TNF)-alpha inhibitors, rifampin, rifabutin, pyrazinamide, isoniazid, ganciclovir or hydroxyurea within 14 days prior to study entry.
* Previous use of any HCV protease or polymerase inhibitor.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would have interfered with adherence to study requirements.
* Serious illness requiring systemic treatment and/or hospitalization within 42 days prior to entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adeel A Butt, MD, MS, Study Chair — University of Pittsburgh; Kenneth E Sherman, MD, PhD, Study Chair — University of Cincinnati CRS
Locations (43):
- United States (42):
  - Alabama CRS, Birmingham, Alabama
  - University of Southern California CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Harbor-UCLA CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Rush University CRS, Chicago, Illinois
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Wayne State Univ. CRS, Detroit, Michigan
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Trinity Health and Wellness Center CRS, Dallas, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - Virginia Commonwealth University CRS, Richmond, Virginia
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Shire NJ, Welge JA, Sherman KE. Response rates to pegylated interferon and ribavirin in HCV/HIV coinfection: a research synthesis. J Viral Hepat. 2007 Apr;14(4):239-48. doi: 10.1111/j.1365-2893.2006.00824.x. PMID 17381715
- [Background] Kwo PY, Lawitz EJ, McCone J, Schiff ER, Vierling JM, Pound D, Davis MN, Galati JS, Gordon SC, Ravendhran N, Rossaro L, Anderson FH, Jacobson IM, Rubin R, Koury K, Pedicone LD, Brass CA, Chaudhri E, Albrecht JK; SPRINT-1 investigators. Efficacy of boceprevir, an NS3 protease inhibitor, in combination with peginterferon alfa-2b and ribavirin in treatment-naive patients with genotype 1 hepatitis C infection (SPRINT-1): an open-label, randomised, multicentre phase 2 trial. Lancet. 2010 Aug 28;376(9742):705-16. doi: 10.1016/S0140-6736(10)60934-8. Epub 2010 Aug 6. PMID 20692693
- [Background] The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009).
- [Result] Sherman KE, Kang M, Sterling R, Umbleja T, Marks K, Alston-Smith B, Greaves W, Butt A. BIRTH: A Phase 3 Trial of Boceprevir/Pegylated Interferon/Ribavirin in HCV/HIV. IDWeek. San Diego, CA. October, 2015. [Abstract 903]

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from May 2012 to December 2013 at 42 U.S. sites.
Groups:
- HCV Treatment-Naive (Group A): Participants were prescribed a lead-in with PEG-IFN and RBV for 4 weeks. After the lead-in, BOC was added. Cirrhotic participants received 44 weeks of triple therapy (BOC+PEG-IFN+RBV). Among non-cirrhotics, the week 8 serum HCV RNA was used to determine total duration of therapy. Those who had undetectable HCV RNA at Week 8 completed therapy at Week 28. Those with detectable HCV RNA at Week 8 received 32 weeks of triple therapy followed by 12 additional weeks of PEG-IFN+RBV.
Period: Overall Study
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Started | 135 | 127
Completed | 81 | 78
Not Completed | 54 | 49
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Lost to Follow-up | 12 | 6
Not completed — Adverse Event | 0 | 3
Not completed — Site closure | 22 | 14
Not completed — Non-adherence to study requirements | 4 | 7
Not completed — Alternate HCV treatment | 7 | 8
Not completed — Ineligible | 0 | 5
Not completed — Nurse error | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants enrolled (Group B participants who were found ineligible after enrollment, n=5, were excluded).
Groups:
- Total: Total of all reporting groups
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B) | Total
Number analyzed (Participants) | 135 | 122 | 257
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [44 to 57] | 53 [49 to 57] | 52 [47 to 57]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at birth.
  Participants
    Female | 25 | 29 | 54
    Male | 110 | 93 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 28 | 45
  Not Hispanic or Latino | 117 | 93 | 210
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 73 | 53 | 126
  White | 57 | 58 | 115
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 135 | 122 | 257
Intravenous Drug Use History [Number; unit: participants]
  Never | 71 | 70 | 141
  Previously | 64 | 52 | 116
Cirrhosis Status at Screening [Number; unit: participants] — Liver cirrhosis was defined as cirrhosis identified by screening liver biopsy or screening FibroSure score greater than 0.74.
  participants
    Cirrhotic | 18 | 38 | 56
    Non-cirrhotic | 117 | 84 | 201
HCV RNA at Entry [Median (Inter-Quartile Range); unit: log10 IU/mL] — Group A: Among n=134 participants with samples collected.
  log10 IU/mL | 6.7 [6.2 to 7.1] | 6.9 [6.5 to 7.3] | 6.8 [6.4 to 7.2]
ART Regimen at Entry [Number; unit: participants]
  EFV + 2 NRTIs | 58 | 51 | 109
  RAL + 2 NRTIs | 47 | 45 | 92
  LPV/RTV + 2 NRTIs | 4 | 4 | 8
  ATV/RTV + 2 NRTIs | 18 | 10 | 28
  DRV/RTV + 2 NRTIs | 6 | 6 | 12
  Not on ART | 2 | 6 | 8
CD4 Cell Count at Entry [Median (Inter-Quartile Range); unit: cells/mm^3] — Among n=133 Group A and n=120 Group B participants who had results available.
  cells/mm^3 | 646 [462 to 818] | 622 [489 to 859] | 625 [473 to 835]
HIV-1 RNA Quantitation at Entry [Number; unit: participants] — Unquantifiable HIV-1 RNA was defined as below the lower limit of the assay (LLOQ). Abbott RealTime HIV-1 assay (LLOQ=40 copies/ml) or Roche COBAS Ampliprep/Taqman HIV-1 assay (LLOQ=20 copies/ml) was used.
  participants
    Unquantifiable | 133 | 113 | 246
    Quantifiable | 0 | 9 | 9
    Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at 24 Weeks After Treatment Discontinuation (SVR24)
Description: SVR24 was defined as undetectable HCV RNA (below the lower limit of quantitation of the assay and target not detected by Roche COBAS® TaqMan® HCV Test v2.0) at 24 weeks after treatment discontinuation. Participants without HCV RNA for SVR24 determination were considered not to have achieved SVR24.
Time Frame: 24 weeks after treatment discontinuation
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Number analyzed (Participants) | 135 | 122
percentage of participants | 34.8 [27.3 to 43.2] | 25.4 [18.5 to 33.8]

2. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events (AEs)
Description: Number of participants who experienced an AE (sign or symptom or laboratory abnormality) of Grade 3 or higher at any time after baseline while on study. The AEs were graded by the clinicians according to the Division of AIDS (DAIDS) AE Grading Table (see references in the Protocol Section) as follows: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening.
Time Frame: From study treatment dispensation to Week 72
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Number analyzed (Participants) | 135 | 122
percentage of participants | 74.1 [66.1 to 80.7] | 73.8 [65.3 to 80.8]

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 12 Weeks After Treatment Discontinuation (SVR12)
Description: SVR12 was defined as undetectable HCV RNA (below the lower limit of quantitation of the assay and target not detected by Roche COBAS® TaqMan® HCV Test v2.0) at 12 weeks after treatment discontinuation. Participants without HCV RNA for SVR12 determination were considered not to have achieved SVR12.
Time Frame: 12 weeks after treatment discontinuation
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Number analyzed (Participants) | 135 | 122
percentage of participants | 35.6 [28.0 to 43.9] | 30.3 [22.9 to 39.0]

4. Secondary Outcome: Percentage of Participants With HIV-1 Viral Load <50 Copies/mL
Description: HIV-1 RNA testing was performed with Abbott RealTime HIV-1 assay (LLOQ=40 copies/mL) or with Roche COBAS AmpliPrep/Taqman HIV-1 assay (LLOQ=20 copies/mL).
Time Frame: Entry and weeks (W) 4, 8, 12, 24, 28, 40, 48, 52, 60, 72
Population: All eligible participants with HIV-1 RNA result available at the respective visit (numbers of participants in Category Titles below; n). Participants who discontinued treatment early due to HCV virologic failure, safety or any other reason started following a separate visit schedule and are not included here.
Measure: Number; unit: percentage of participants
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Number analyzed (Participants) | 135 | 122
percentage of participants
  W0 HIV-1 RNA (A: n=133, B: n=122) | 100.0 | 92.6
  W4 HIV-1 RNA (A: n=123, B: n=114) | 98.4 | 96.5
  W8 HIV-1 RNA (A: n=117, B: n=104) | 100.0 | 96.2
  W12 HIV-1 RNA (A: n=108, B: n=99) | 98.1 | 98.0
  W24 HIV-1 RNA (A: n=62, B: n=52) | 100.0 | 100.0
  W28 HIV-1 RNA: (A: n=54, B: n=45) | 98.1 | 100.0
  W40 HIV-1 RNA (A: n=52, B: n=38) | 92.3 | 100.0
  W48 HIV-1 RNA (A: n=23, B: n=33) | 100.0 | 100.0
  W52 HIV-1 RNA (A: n=24, B: n=0) | 100.0 | NA — Group B participants did not have a study visit at Week 52.
  W60 HIV-1 RNA (A: n=40, B: n=36) | 100.0 | 97.2
  W72 HIV-1 RNA (A: n=34, B: n=27) | 97.1 | 100.0

5. Secondary Outcome: CD4+ T-Cell Count (CD4) Change From Baseline
Description: Change in CD4 T-cell count was calculated as value at the post entry visit minus the value at entry.
Time Frame: Entry and weeks (W) 8, 12, 24, 28, 40, 48, 52, 60, 72
Population: All eligible participants enrolled with CD4 result available from entry and the respective post-entry visit (numbers of participants in Category Titles below; n). Participants who discontinued treatment early due to HCV virologic failure, safety or any other reason started following a separate visit schedule and are not included here.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Number analyzed (Participants) | 135 | 122
cells/mm^3
  W8 CD4 change (A: n=115, B: n=101) | -174 [-285 to -77] | -170 [-290 to -83]
  W12 CD4 change (A: n=106, B: n=95) | -194 [-342 to -101] | -202 [-331 to -90]
  W24 CD4 change (A: n=61, B: n=52) | -277 [-402 to -143] | -263 [-418 to -184]
  W28 CD4 change (A: n=53, B: n=44) | -304 [-441 to -157] | -284 [-412 to -227]
  W40 CD4 change (A: n=50, B: n=37) | -128 [-234 to -47] | -276 [-368 to -180]
  W48 CD4 change (A: n=22, B: n=35) | -220 [-420 to -77] | -237 [-352 to -147]
  W52 CD4 change (A: n=23, B: n=0) | -24 [-174 to 75] | NA [NA to NA] — Group B participants did not have a study visit at Week 52.
  W60 CD4 change (A: n=39, B: n=36) | -34 [-210 to 107] | -79 [-146 to 40]
  W72 CD4 change (A: n=33, B: n=27) | 8 [-123 to 77] | -15 [-129 to 124]

6. Secondary Outcome: Number of Participants With Undetectable HCV RNA at Week 4, 8 and 12 Study Visits
Description: Undetectable HCV RNA was defined as below the lower limit of quantitation of the assay and target not detected by Roche COBAS® TaqMan® HCV Test v2.0.
Time Frame: Weeks (W) 4, 8, 12
Population: All eligible participants with HCV RNA result available at the respective visit (numbers of participants in Category Titles below; n). Participants who discontinued treatment early due to HCV virologic failure, safety or any other reason started following a separate visit schedule and are not included here.
Measure: Number; unit: participants
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Number analyzed (Participants) | 135 | 122
participants
  W4 HCV RNA (A: n=122, B: n=116) | 9 | 3
  W8 HCV RNA (A: n=117, B: n=104) | 48 | 28
  W12 HCV RNA (A: n=109, B: n=99) | 68 | 43

7. Secondary Outcome: Number of Participants With Undetectable HCV RNA at Week 16, 20, 24 and 28 Study Visits
Description: Undetectable HCV RNA was defined as below the lower limit of quantitation of the assay and target not detected by Roche COBAS® TaqMan® HCV Test v2.0. This outcome measure was intended for a potential interim analysis when study data up to Week 28 were complete. However, this interim analysis was not conducted.
Time Frame: Weeks (W) 16, 20, 24, and 28
Population: This outcome measure was intended for a potential interim analysis which was not conducted.
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Grade 2 or Higher Signs and Symptoms and Laboratory Abnormalities and Other Serious AEs
Description: This outcome measure was intended for a potential interim analysis when study data up to Week 28 were complete. However, this interim analysis was not conducted. Refer to Outcome Measure 2 above for the safety outcome that includes the whole study duration from entry to week 72.
Time Frame: From study treatment dispensation to Week 28
Population: This outcome measure was intended for a potential interim analysis which was not conducted.
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From study treatment dispensation to Week 72.
Description: The protocol required reporting of signs/symptoms >=Grade 2, laboratory results >=Grade 3 and events that led to a change in treatment, regardless of grade. HGB, PLT, ANC, AST, ALT, INR, total and direct bilirubin, creatinine were reported regardless of grade. The DAIDS AE Grading Table (V1.0) and Expedited AE Manual (V2.0) were used.
Arm/Group | HCV Treatment-Naive (Group A) | HCV Treatment-Experienced (Group B)
Serious Adverse Events (participants affected / at risk) | 32/135 | 31/122
Other Adverse Events (participants affected / at risk) | 135/135 | 120/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HCV Treatment-Naive (Group A) (N=135) | HCV Treatment-Experienced (Group B) (N=122)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 9
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 2 | 0
Injection site mass (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Liver disorder (Hepatobiliary disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Injection site cellulitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Perinephric abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Toxoplasmosis (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 3 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Lipase increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Priapism (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HCV Treatment-Naive (Group A) (N=135) | HCV Treatment-Experienced (Group B) (N=122)
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Diarrhoea (Gastrointestinal disorders) | 9 | 13
Nausea (Gastrointestinal disorders) | 28 | 28
Vomiting (Gastrointestinal disorders) | 18 | 13
Asthenia (General disorders) | 3 | 7
Chills (General disorders) | 17 | 16
Fatigue (General disorders) | 44 | 34
Malaise (General disorders) | 7 | 7
Pain (General disorders) | 4 | 8
Pyrexia (General disorders) | 13 | 12
Alanine aminotransferase increased (Investigations) | 72 | 66
Aspartate aminotransferase increased (Investigations) | 95 | 89
Blood albumin decreased (Investigations) | 8 | 6
Blood alkaline phosphatase increased (Investigations) | 10 | 18
Blood bicarbonate decreased (Investigations) | 13 | 10
Blood bilirubin increased (Investigations) | 32 | 37
Blood creatinine increased (Investigations) | 27 | 21
Blood glucose decreased (Investigations) | 11 | 4
Blood glucose increased (Investigations) | 26 | 29
Blood phosphorus decreased (Investigations) | 10 | 9
Blood potassium decreased (Investigations) | 9 | 9
Blood sodium decreased (Investigations) | 11 | 14
Blood uric acid increased (Investigations) | 11 | 21
Haemoglobin decreased (Investigations) | 74 | 68
Lipase abnormal (Investigations) | 12 | 20
Lipase increased (Investigations) | 6 | 12
Neutrophil count decreased (Investigations) | 115 | 95
Platelet count decreased (Investigations) | 68 | 73
Weight decreased (Investigations) | 20 | 26
White blood cell count decreased (Investigations) | 35 | 34
Decreased appetite (Metabolism and nutrition disorders) | 16 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 13
Dizziness (Nervous system disorders) | 7 | 9
Headache (Nervous system disorders) | 13 | 16
Anxiety (Psychiatric disorders) | 10 | 5
Depression (Psychiatric disorders) | 10 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Erythema (Skin and subcutaneous tissue disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less